CLINICAL TRIAL: NCT00179894
Title: Improving Medication Use for ADHD in Primary Care
Brief Title: Improving Attention Deficit Hyperactivity Disorder Treatment Adherence and Outcome in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John V. Lavigne, Chief Psychologist, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01MH066866 (NIH); R01MH066866 (NIH); DSIR 82-SECH
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Physician training (Experimental): Physician participants will receive training in guidelines and medication monitoring
  Interventions: Behavioral: Physician training
- 2 (No Intervention): Physician participants will provide usual care and no special intervention

INTERVENTIONS:
Behavioral: Physician training — Physicians are trained in guidelines for medication management.
  Arms: 1 Physician training

SUMMARY:
This study will determine the effectiveness of educating pediatricians about attention deficit hyperactivity disorder treatment guidelines in improving child behavior and pediatricians' adherence to medication guidelines.

DETAILED DESCRIPTION:
The most effective treatment for improving the core symptoms of inattention, impulsivity and hyperactivity in children with attention deficit hyperactivity disorder (ADHD) involves the use of stimulant medications. Most children with ADHD are treated by pediatricians, but the treatment provided is often less than optimal. This study is designed to see if training for pediatricians in following guidelines for management of first-line medicines for ADHD leads to improvement in child behavior, and whether the physicians can adhere to the guidelines.

Over 100 studies have shown that stimulant medications are effective for improving the core symptoms of Attention Deficit Hyperactivity Disorder (ADHD). Approximately 70% of children who receive ADHD medications are treated by their primary care pediatrician, but studies show that management is not always optimal. The present study is designed to see if child behavior can be improved by training pediatricians in the use of guidelines for treating ADHD, and whether the physicians can adhere to the guidelines. Twenty-four pediatric practices were randomized to a treatment as usual or specialized care (receiving training in guidelines and computer assisted monitoring of patient progress and medication titration). Children are assessed with parent and teacher reports at baseline, 4-, 9-, and 12-months post initiation of treatment, and classroom observations of behavior are assessed at baseline, 6-, and 12-months. Approximately 400 children are to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ADHD
* Not currently on medication

Exclusion Criteria:

* No serious neurological disorders of sever mental health problems (suicidal behavior, autism)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2003-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Behavior changes as rated by teachers | Measured at Month 12

SECONDARY OUTCOMES:
Behavior change as rated by parents | Measured at Month 12
Behavior changes as rated by classroom observation | Measured at Month 12
Relation between adherence to protocol and behavior change | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: John V. Lavigne, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States